CLINICAL TRIAL: NCT03868527
Title: The ARCAN Database is Used for Retrospective Non-interventional Research Projects. The Database Collects Clinical and Laboratory Data From Patients With Lymphoid Malignancies. The Database Doesn't Require Biological Sample of Patients, it Records Only Information Based on the Patients' Medical File.
Acronym: Arcan database
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ARCAN Database
Record Dates: First submitted 2019-02-26; First posted 2019-03-11 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematological diseases: Cohort of patients followed for lymphoid malignant hemopathy in Lyon Sud Hospital
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Data collection for biostatistical analysis about hematological diseases

SUMMARY:
To identify the diagnostic and therapeutic approach (efficacy and toxicity) of patients with lymphoid malignant hemopathy who are managed in the hematology department.

ELIGIBILITY:
Inclusion Criteria:

- Patients followed for hematological diseases in Lyon Sud Hospital

Exclusion Criteria:

- Patients who doesn't have hematological diseases

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed for lymphoid malignant hemopathy in Lyon Sud Hospital
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2003-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 730 days
  Period between the end of the first treatment and the first confirmed relapse of lymphoma of patients who have received treatment to treat their lymphoma.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Salles, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France